CLINICAL TRIAL: NCT05357261
Title: Deliver-EE: Evaluating Effects of Meal Delivery on the Ability of Homebound Older Adults to Remain in the Community Via A Pragmatic, Two-Arm, Randomized Comparative Effectiveness Trial
Brief Title: Deliver-EE: Evaluating Effects of Meal Delivery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Meals on Wheels America (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022003287; IHS-2020C3-21201 (Other Grant/Funding Number: Patient-Centered Outcomes Research Institute)
Record Dates: First submitted 2022-04-27; First posted 2022-05-02 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Healthy
Keywords: Homebound; Nutrition; Food insecurity
MeSH Terms: interventions — Fast Foods

STUDY DESIGN:
Intervention Model Description: To evaluate the effectiveness of receiving daily-delivered meals with a wellness check and socialization versus frozen, drop-shipped meals on food insecure, homebound older adults' ability to remain in the community and out of institutional settings.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Daily home delivered meals (Active Comparator): A lunch-time meal delivered to participants' homes five days per week with wellness check and socialization.
  Interventions: Behavioral: Wellness Check and Socialization; Other: Prepared Meals
- Frozen, Drop-shipped Meals (Experimental): Ten frozen meals that are mailed to participants every two weeks.
  Interventions: Other: Prepared Meals

INTERVENTIONS:
Behavioral: Wellness Check and Socialization — In-home delivery with opportunity for driver observation and interaction
  Arms: Daily home delivered meals
Other: Prepared Meals — Prepared meals compliant with Older Americans Act nutrition programs guidelines

SUMMARY:
This study will randomly assign 2,300 older adults on waiting lists at fourteen Meals on Wheels programs in Florida, Illinois, Maryland, Tennessee, Texas, North Carolina, South Carolina, and California into two groups who will receive: (a) daily delivery of meals, five days a week or (b) a shipment of 10 frozen meals, every two weeks. Researchers will examine participants' Medicare claims to understand if differences in healthcare utilization occur between the two groups within six months after they start receiving meals. Researchers will also ask participants questions prior to receiving meals, and again at three months, to understand how meals impact their ability to obtain food, their feelings of loneliness, and their overall quality of life. The primary study outcome will be the ratio of days spent in institutional settings (i.e., hospital, nursing home) in the six months after participants begin receiving meals. The secondary outcomes include the ratio of days spent in institutional settings in the three months after participants begin receiving meals, food insecurity, subjective isolation/loneliness, and health-related quality of life. The team will also examine differences in dietary intake between the two groups as an exploratory outcome.

DETAILED DESCRIPTION:
Background and Significance: Food insecurity among older adults is a critical public health issue with implications for families, the healthcare system, and society. In 2017, an estimated 5.5 million older adults (7.7%) in the United States were food insecure. Among older adults, food insecurity is associated with poor health status and outcomes and accounts for an estimated $130 billion annually in medical expenses. As a result, healthcare entities (e.g., payers, integrated systems, providers) are increasingly interested in addressing food insecurity, among other social risk factors, through non-medical services such as home-delivered meals to older patients and enrollees. Home-delivered meals, long provided through a network of community-based organizations funded through the Older Americans Act, state dollars, and charitable contributions, promote food security, socialization, and independence among older adults. While meals have traditionally been provided daily to clients' homes by a volunteer or paid driver, mailed frozen meals have emerged in recent years as a lower cost alternative. However, there is limited evidence about what mode of delivery is most effective in promoting community independence, reducing healthcare utilization, and improving patients' quality of life, as well as how these outcomes may vary as a function of patients' preferences for how meals are delivered to them.

Study Aims: The long-term goal of this research is to generate evidence to guide patient, family, meal programs, and healthcare entities' decision-making about which mode of meal delivery is best for promoting important, patient-centered outcomes. This will be accomplished through three specific aims: 1) To evaluate the effectiveness of receiving daily-delivered meals with a safety check and socialization versus frozen, drop-shipped meals on food insecure, homebound older adults' ability to remain in the community; 2) To understand food insecure, homebound older adults' preferences for mode of meal delivery and the effect of receiving a meal that is concordant with their preference on their ability to remain in the community; and 3) To measure and quantify secondary outcomes prioritized by stakeholders related to these different modes of meal delivery.

Study Description: This is a two-arm pragmatic, randomized controlled trial that will compare participants' health outcomes between two conventional approaches for delivering meals to food insecure, homebound older adults at thirteen diverse Meals on Wheels America member programs in Florida, Illinois, Maryland, Tennessee, Texas, California, North Carolina, and South Carolina. The comparators are the two main modes of meal delivery used in everyday practice: daily-delivered meals and drop-shipped, frozen meals. A total of 2300 food insecure, homebound older adults (ages 66+) on waiting lists at these programs will be enrolled in the study; 1150 older adults will receive meals delivered five days per week, with socialization and a wellness check by a volunteer or paid driver, and 1150 will receive a box of 10 frozen meals that will be mailed to participants every two weeks. The primary outcome will be the ratio of days that a participant is in an institutional setting (i.e., hospital, nursing home) in the six months following the start of meal delivery and will be derived from data from the Centers for Medicare and Medicaid Services; secondary outcomes include the ratio of days in institutional settings in the three months following the start of meal delivery, food insecurity, loneliness, and quality of life. Secondary outcomes will be derived from Centers for Medicare and Medicaid Services' data and surveys with participants. Self-reported dietary intake will be included as an exploratory outcome. To examine heterogeneity of treatment effects, the investigators will test for interactions between the two types of meals and participants' preferences for meals, as well as clients' living arrangements. This research will be the first to prospectively evaluate the comparative effectiveness of the two predominant meal delivery options in partnership with a variety of stakeholders. The knowledge generated from this research will be of tremendous value to healthcare payers, health systems, providers, community-based organizations, patients, and their families, because it will identify the mode of meal delivery that best meets older, homebound, and food insecure patients' needs and promotes community independence

ELIGIBILITY:
Inclusion Criteria:

* Age 66+
* On program waiting list
* Must reside in program's daily service area
* Must be able to eat a general diet with no dietary restrictions

Exclusion Criteria:

* Primary language is not English or Spanish
* Has end stage renal disease/requires specialized renal diet
* Unable to participate in a phone survey/interview (e.g., difficulty hearing, lack of comprehension of study purpose, does not have working phone)

Min Age: 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 2300 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
6-Month Ratio of Days in Institutional Settings | 6 months
  Ratio between the number of days that are spent in an institutional setting (i.e., acute care hospital, psychiatric hospital, long-term care hospital, nursing home, or skilled nursing facility) and the number of days alive in the six months following receipt of meals

SECONDARY OUTCOMES:
3-Month Ratio of Days in Institutional Settings | 3 months
  Defined similarly to the primary outcome, but assesses the immediate (3-month) impact of meals on days spent in institutional settings
Food Insecurity | 3 months
  U.S. Household Food Security Survey Module: Six-Item Short Form; Minimum value (0) indicates high food insecurity; Maximum value (6) indicates very low food insecurity
Subjective Isolation/Loneliness | 3 months
  University of California, Los Angeles 3-Item Loneliness Scale; Minimum value (3) indicates low feelings of loneliness; Maximum value (9) indicates high feelings of loneliness
Health-Related Quality of Life | 3 months
  The Centers for Disease Control and Prevention's Health-Related Quality of Life 4-question core modules, called the "Healthy Days Measures"; The unhealthy days index is calculated by summing the number of physically and mentally unhealthy days, capped at 30 total days.

CONTACTS AND LOCATIONS:
Overall Officials: Kali S. Thomas, PhD, Principal Investigator — Johns Hopkins University School of Nursing; Kimberly P. Bernard, PhD, Principal Investigator — Brown University School of Public Health
Locations (14):
- United States (14):
  - Meals on Wheels San Diego County, San Diego, California
  - Neighborly Care Network, Clearwater, Florida
  - Aging True, Jacksonville, Florida
  - Meals on Wheels Northeastern Illinois, Evanston, Illinois
  - Meals on Wheels of Central Maryland, Baltimore, Maryland
  - Meals On Wheels Durham, Durham, North Carolina
  - Senior Resources of Guilford, Greensboro, North Carolina
  - Meals On Wheels - Anderson, Anderson, South Carolina
  - Senior Resources Inc, Columbia, South Carolina
  - Metropolitan Inter-Faith Association (MIFA), Memphis, Tennessee
  - Visiting Nurse Association of Texas, Dallas, Texas
  - Northwest Assistance Ministries, Houston, Texas
  - Amigos Del Valle, Inc, Mission, Texas
  - Meals on Wheels San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thomas KS, Bernard KP, Clark M, Dionne L, Fisher A, Gadbois E, Harrison J, Juckett L, Locher J, Risica P, Sequeira T, Theilheimer L, Gutman R. Evaluating effects of meal delivery on the ability of homebound older adults to remain in the community via a pragmatic, two-arm, randomized comparative effectiveness trial: study protocol for the Deliver-EE trial. Trials. 2024 Nov 22;25(1):787. doi: 10.1186/s13063-024-08635-3. PMID 39574158
- [Derived] Juckett LA, Bernard KP, Clark MA, Gadbois EA, Wright B, Thomas KS. Core functions and forms in home-delivered meal programs: a stakeholder-driven approach to identifying essential practices. Implement Sci Commun. 2025 Apr 14;6(1):43. doi: 10.1186/s43058-025-00728-7. PMID 40229891
- [Derived] Juckett LA, Bernard KP, Thomas KS. Partnering with social service staff to implement pragmatic clinical trials: an interim analysis of implementation strategies. Trials. 2023 Nov 17;24(1):739. doi: 10.1186/s13063-023-07757-4. PMID 37978528